CLINICAL TRIAL: NCT01788969
Title: Serotonergic Modulation of Motor Function in Subacute and Chronic SCI
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Thomas G Hornby, Principle Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00014259
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Spinal Cord Injury
Keywords: Gait training; Lexapro; Tizanidine
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gait Training with Lexapro (Experimental): Gait training 2 weeks, gait training 4 weeks (3 X week) with Lexapro (10mg SSRI), wash out period of 1 week, gait training, for 4 weeks with placebo (10 mg). Patients will also be provided prescribed TIZ by their physician to help control of spastic motor behaviors.
  Interventions: Drug: Lexapro
- Gait Training with Placebo (Active Comparator): Gait training 2 weeks, gait training for 4 weeks (3X week) with Placebo (10 mg), wash out period of 1 week, gait training for 4 weeks with Lexapro(10 mg). Patients will also be provided prescribed TIZ by their physician to help control of spastic motor behaviors.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lexapro — Agent + training vs Placebo + training
  Other Names: escitalopram
  Arms: Gait Training with Lexapro
Drug: Placebo — Agent + training vs Placebo + training
  Other Names: microcrystalline dextrose
  Arms: Gait Training with Placebo

SUMMARY:
The manifestation of weakness and involuntary reflexes following motor incomplete spinal cord injury (SCI) may be partly a result of damage to descending pathways to the spinal cord that release serotonin. In models of SCI, for example, application of agents that simulate serotonin has been shown to modulate voluntary motor behaviors, including augmentation of walking recovery. In humans following neurological injury, the effects of 5HT agents are unclear. Few previous reports indicate improved motor function following administration of agents which enhance the available serotonin in the brain, although some data suggests that decreased serotonin may be beneficial. In this application, the investigators propose to study the effects of clinically used agents that increase or decrease intrinsic serotonin activity in the brain on strength and walking ability following human motor incomplete SCI. Using detailed electrophysiological recordings, and biomechanical and behavioral measures, the investigators will determine the effects of acute or chronic doses of these drugs on voluntary and involuntary motor behaviors during static and dynamic conditions. The novelty of this proposed research is the expectation that agents that enhance serotonin activity may increase abnormal reflexes in SCI, but simultaneously facilitate motor and walking recovery. Despite potential improvements in voluntary function, the use of pharmacological agents that may enhance spastic motor behaviors following SCI is in marked contrast to the way in which drugs are typically used in the clinical setting.

DETAILED DESCRIPTION:
The proposed study will consist of a double-blinded, randomized controlled trial using a crossover design to assess the effects of SSRIs (escitalopram oxalate, Lexapro®, Forest Pharmaceuticals, Inc) and 5HT-antagonists (cyproheptadine [CYPRO], Periactin ®, Merck, Inc) on volitional and spastic motor behaviors in subjects with motor incomplete SCI following both acute and chronic medication delivery. Voluntary and reflexive motor behaviors in 120 subjects with SCI will be assessed. These interventions will be applied to individuals with acute (< 6 months post injury) chronic (> 1 year post injury) motor incomplete SCI to determine both the rate and extent of changes in volitional motor performance and involuntary spastic behaviors. For the training portion of the study (referred to as subproject 2 below), a portion of the acute and chronic subjects will be evaluated every 2 weeks for up to16 weeks and participate in locomotor training, to investigate and better understand changes in motor function and recovery in individuals with spinal cord injuries. Following 2-4 weeks of this training, individuals will be given either the study drug, or placebo and continue evaluation and training. Following an additional 4 weeks, subjects will be given either the placebo or study drug (whichever they did not receive during the prior 4 weeks). The order will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* age of subjects between 18 and 65 years of age, due to the effects of greater age on functional recovery of ambulation (Penrod et al. 1990);
* medically stable with medical clearance from the subject's primary internist or physiatrist to participate;
* level of the lesion between C5-T10 spinal cord level due to non-progressive etiology;
* <6 months or >1 yr since initial injury. Range of motion requirements include: ankle dorsiflexion ankle to 10 degrees and plantarflexion to 30 degrees, knee flexion from 0 to 120 degrees, hip flexion to 90 degrees, and hip extension to 10 degrees.

Exclusion Criteria:

* presence of concurrent severe medical illness, including unhealed decubiti, existing infection, cardiovascular disease, significant osteoporosis (as indicated by history of fractures following injury)
* active heterotrophic ossification in the lower extremities
* known history of peripheral nerve injury in lower legs
* history of known traumatic head injury
* a history of cardiovascular or pulmonary complications, including significant obstructive and/or restrictive lung diseases
* inability to tolerate 30 minutes of standing without orthostasis (decrease in blood pressure by 20 mmHg systolic and 10 mmHg diastolic)
* individuals who are undergoing concurrent physical therapy will be excluded to eliminate confounding effects
* women of childbearing potential will not be excluded, although women who are pregnant will be excluded due to the lack of proven safety of pharmacological agents in pregnant women
* cranial stimulation exclusions: history of epilepsy or a seizure event, metal implants in the head or face, unexplained and recurring headaches, skull abnormalities or fractures, implanted cardiac pacemaker or suffered a concussion within the last 6 months
* interactions with other medications or previous sensitivity to SSRIs, 5-HT antagonists or anti-histamines
* patients prescribed medications for alleviation of spastic motor behaviors, anti-depressant medications, or other medications with known interactions to SSRIs will be excluded from participation unless both attending physician and patient agree to cease all such medications during the evaluation and training period. A 14-day minimum washout period for all such medications will be utilized
* patients with known liver, renal, or other metabolic disease that may interfere with drug action and/or clearance will be excluded from the proposed study. The low daily dosage of the agent to be used (10 mg Lexapro and 16 mg Cypro) has shown very little side effects with patients with hepatic or renal disease
* patients who are diagnosed or previously diagnosed with depression will be excluded. A preliminary screening tool (Center for Epidemiological Studies - Depression Scale) will be administered to all patients. Scores > 16 indicate symptoms of depression. For those patients, a physician will be required to evaluate the subject to determine eligibility.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-06; Primary Completion 2016-12 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Walking Index for Spinal Cord Injury (WISCI II) | Compare changes in WISCI II pre to post training with placebo to pre to post training with Lexapro during a 10-12 week time period.
  Evaluation of bracing, assistive device, and assistance required for ambulation

SECONDARY OUTCOMES:
Volitional Strength | Pre Training (Day 1), Pre Drug B (approx end of week 5), Post Final (approx end of week 10)
  Ankle, knee, hip flexors/extensors strength (Nm) tested bilaterally (Biodex®)
Gait kinematics | Pre Training (Day 1), Pre Drug A (approx end of week 2), Post Drug A (approx end of week 4), Pre Drug B (approx end of week 5), Post Drug B (approx end of week 9), Post-Final (approx end of week 10)
  Kinematic excursions of hip/knee/ankle (Motion Analysis®)
Fastest possible walking velocity over ground (FV; m/s) | Pre Training (Day 1), Pre Drug A (approx end of week 2), Post Drug A (approx end of week 4), Pre Drug B (approx end of week 5), Post Drug B (approx end of week 9), Post-Final (approx end of week 10)
  Subject walks a distance of 10m with the middle 6m being timed. Instructions to walk normal comfortable pace.
Six minute walking distance (m) | Pre Training (Day 1), Pre Drug A (approx end of week 2), Post Drug A (approx end of week 4), Pre Drug B (approx end of week 5), Post Drug B (approx end of week 9), Post-Final (approx end of week 10)
  Subject asked to walk normal comfortable pace for 6 minutes. Total distance is recorded. Subject can take rest breaks as needed but are encouraged to continue walking throughout the 6 minutes.
Lower Extremity Motor Scores (LEMS) | Pre Training (Day 1), Pre Drug A (approx end of week 2), Post Drug A (approx end of week 4), Pre Drug B (approx end of week 5), Post Drug B (approx end of week 9), Post-Final (approx end of week 10)
  Measure of lower extremity muscle strength on 0-5 point scale
Modified Ashworth of knee extensors/flexors (ModAsh) | Pre Training (Day 1), Pre Drug A (approx end of week 2), Post Drug A (approx end of week 4), Pre Drug B (approx end of week 5), Post Drug B (approx end of week 9), Post-Final (approx end of week 10)
  Measure of spasticity of knee flexors and extensors during passive range of motion
Spinal Cord Assessment Tool for Spasticity (SCATS) | Pre Training (Day 1), Pre Drug A (approx end of week 2), Post Drug A (approx end of week 4), Pre Drug B (approx end of week 5), Post Drug B (approx end of week 9), Post-Final (approx end of week 10)
  Measure of spasticity tested in supine
Peak Treadmill Velocity | Compare changes in peak treadmill velocity pre to post training with placebo to pre to post training with Lexapro during a 10-12 week time period.
  Peak treadmill speed during graded treadmill testing

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G Hornby, PhD, PT, Principal Investigator — Rehabiltiation Institute of Chicago/UIC
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States